CLINICAL TRIAL: NCT02452983
Title: SS1: Pilot Study of Sertraline in Treatment of Low-Risk Myelodysplastic Syndrome (MDS)
Brief Title: Sertraline in Treatment of Low-Risk Myelodysplastic Syndrome
Acronym: SS1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This protocol is closed to further enrollment due to lack of study progress.
Sponsor: Gustavo Rivero (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Gustavo Rivero, Assistant Professor, Principal Investigator, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-36160
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Myelodysplastic Syndromes
Keywords: Anemia; Leukemia; Hematologic diseases; Cytopenias; Bone marrow diseases; Preleukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia; Leukemia; Hematologic Diseases; Cytopenia; Bone Marrow Diseases; Preleukemia | interventions — Sertraline; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sertraline (Experimental): Sertraline tablets 100mg daily for 4 (28-day) cycles
  Interventions: Drug: Sertraline; Procedure: Bone Marrow Aspirate/Biopsy

INTERVENTIONS:
Drug: Sertraline
  Other Names: Zoloft
Procedure: Bone Marrow Aspirate/Biopsy

SUMMARY:
This study will investigate the effects of sertraline in people with low-risk myelodysplastic syndrome (MDS). It is hoped that sertraline will decrease disease progression and reduce the need for blood transfusions.

DETAILED DESCRIPTION:
This pilot study investigates clinical benefit of four 28-day cycles of sertraline in low-risk MDS patients. Participants will receive 100mg of oral sertraline daily. The study will also evaluate potential associated biological mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Very Low or Low risk MDS defined by IPSS-R confirmed by a bone marrow aspirate and biopsy (Blast count must be < 20%)
* Hemoglobin < 11 g/dL, or transfusion dependency.
* Platelet count <100,000/mm3
* Absolute Neutrophil Count (ANC) < 1000/mm3
* Life expectancy of 12 months or greater
* ECOG Performance status of 0 - 3
* Age ≥ 18 years
* Willing to use medically acceptable methods of birth control during the study and for 28 days after discontinuing study treatment
* All subjects must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* Both men and women and members of all races and ethnic groups

Exclusion Criteria:

* Previous exposure to 5-AC (azacitidine) or decitabine
* Use of antidepressants such as sertraline within 6 weeks OR use of paroxetine, fluoxetine, or citalopram within 3 months prior to registration
* Active cases (within past 12 months) of depressive disorder, manic episodes, and/or anxiety requiring active treatment with an SSRI. Patients being treated with an SSRI for non-psychiatric indication are allowed, and should go through the appropriate washout.
* Previous or concurrent malignancy, except treated basal cell or squamous cell cancer of skin, treated in situ cervical cancer, treated lobular or ductal carcinoma in situ in one breast, or any other cancer for which the patient has been disease-free for at least 5 years
* Actively receiving chemo-immunotherapy
* Evidence of active infection
* Treatment with steroids or immunosuppressive therapy such as cyclosporine, tacrolimus, anti-thymocyte globulin (ATG) within 6 months of registration
* Platelet transfusion within 8 weeks of registration.
* Platelet count < 20,000/mm3 within 14 days of registration.
* Active treatment with growth factors such erythropoietin stimulating agent (ESA), granulocyte colony-stimulating factor (GCSF), thrombopoietin stimulating factor within 8 weeks of registration
* Treatment with an investigational agent within 4 weeks of registration
* History of autoimmune disease including rheumatoid arthritis, systemic lupus and sarcoidosis
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sertraline
* Known history of splenomegaly
* Pregnant or nursing women are excluded from this study because Sertraline is a Class C agent with the potential for teratogenic or abortive effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sertraline, breast feeding should be discontinued.
* HIV: Given high risk for Immune thrombocytopenic purpura, HIV associated neutropenia and combination antiretroviral therapy, patients with known HIV are excluded because of the potential for pharmacokinetic interactions with sertraline.
* Any condition or illness that, in the Investigator's opinion, would place the subject at unacceptable risk if he/she were to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-05; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Hematological Improvement - minor (HI-minor) | 16 weeks
  Improvement in erythroid, neutrophil or platelet

SECONDARY OUTCOMES:
HI-minor response rate | 4 weeks
  HI-minor response rate Cycle 1
HI-minor response rate | 8 weeks
  HI-minor response rate Cycle 2
HI-minor response rate | 12 weeks
  HI-minor response rate Cycle 3
HI-minor response rate | 16 weeks
  HI-minor response rate Cycle 4
Individual rates of HI minor measurements: erythroid, neutrophil and platelet | 4 weeks
  Individual rates of HI minor measurements at Cycle 1: erythroid, neutrophil and platelet
Individual rates of HI minor measurements: erythroid, neutrophil and platelet | 8 weeks
  Individual rates of HI minor measurements at Cycle 2: erythroid, neutrophil and platelet
Individual rates of HI minor measurements: erythroid, neutrophil and platelet | 12 weeks
  Individual rates of HI minor measurements at Cycle 3: erythroid, neutrophil and platelet
Individual rates of HI minor measurements: erythroid, neutrophil and platelet | 16 weeks
  Individual rates of HI minor measurements at Cycle 4: erythroid, neutrophil and platelet
Hematological Improvement - major (HI-major) response rate | 4 weeks
  HI-major response rate at Cycle 1
Hematological Improvement - major (HI-major) response rate | 8 weeks
  HI-major response rate at Cycle 2
Hematological Improvement - major (HI-major) response rate | 12 weeks
  HI-major response rate at Cycle 3
Hematological Improvement - major (HI-major) response rate | 16 weeks
  HI-major response rate at Cycle 4
Individual rates of HI major measurements: erythroid, neutrophil and platelet | 4 weeks
  Individual rates of HI major measurements at Cycle 1: erythroid, neutrophil and platelet
Individual rates of HI major measurements: erythroid, neutrophil and platelet | 8 weeks
  Individual rates of HI major measurements at Cycle 2: erythroid, neutrophil and platelet
Individual rates of HI major measurements: erythroid, neutrophil and platelet | 12 weeks
  Individual rates of HI major measurements at Cycle 3: erythroid, neutrophil and platelet
Individual rates of HI major measurements: erythroid, neutrophil and platelet | 16 weeks
  Individual rates of HI major measurements at Cycle 4: erythroid, neutrophil and platelet
Serum cytokine level modifications | 4 weeks
  Measured as the difference between Week 4 and pre-treatment levels
Serum cytokine level modifications | 8 weeks
  Measured as the difference between Week 8 and pre-treatment levels
Serum cytokine level modifications | 12 weeks
  Measured as the difference between Week 12 and pre-treatment levels
Serum cytokine level modifications | 16 weeks
  Measured as the difference between Week 16 and pre-treatment levels
Changes in the Gene Expression Profile | Between Baseline and Day 14
  Measured as the difference between Day 14 and Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo A Rivero, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas